CLINICAL TRIAL: NCT04420130
Title: Camrelizumab Combined With Ablation and Chemotherapy in Patients With Pancreatic Cancer Liver Metastasis: a Single-arm, Prospective Study
Brief Title: A Trial of Camrelizumab Combined With Ablation and Chemotherapy in Patients With Pancreatic Cancer Liver Metastasis（SHR-1210-HLJ-009）
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to pass ethics committee review
Sponsor: Yanqiao Zhang (Other)
Responsible Party: Sponsor-Investigator, Yanqiao Zhang, Director of the hospital, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-HLJ-009
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer; Liver Metastasis
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — camrelizumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combined with ablation and chemotherapy (Experimental): First, patients with liver metastases from pancreatic cancer are given ablation of liver metastases, and conventional chemotherapy plus camrelizumab is performed 1 week after surgery. If patients have multiple metastases, ablation treatment needs to be performed in stages, each ablation After 1 week of treatment, sequential chemotherapy + camrelizumab were reinfused, and the efficacy was evaluated every 2 cycles until the disease progressed or the patient could not tolerate it.
  Interventions: Drug: Camrelizumab; Drug: Chemotherapy; Procedure: Ablation

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab was administered 200mg iv every 3 weeks
Drug: Chemotherapy — The chemotherapy regimen may be a standard regimen for routine treatment of advanced pancreatic cancer.
Procedure: Ablation — First give pancreatic cancer patients with liver metastases to ablation of liver metastases

SUMMARY:
This is a a single-arm, prospective study of Camrelizumab combined with ablation and chemotherapy for patients with Pancreatic cancer liver metastasis.

The main purpose of this study is to evaluate the safety and tolerability of Camrelizumab combined with ablation and chemotherapy as a treatment of Pancreatic cancer liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver metastasis of pancreatic cancer diagnosed by histology or cytology;
* Must have CT or MRI examination in the last 3 months;
* With measurable tumor lesions (spiral CT scan ≥10mm, meet RECIST 1.1 standard);
* Expected survival time> 3 months;
* The interval between the end of the patient's previous chemotherapy or adjuvant chemotherapy must be more than 6 months;
* No radiation therapy (unless there is at least one measurable target lesion in the non-irradiated area);
* Must score pain;
* Age: 18 to 70 years old, male or female;
* ECOG PS: 0-1 points;
* The functions of important organs meet the following requirements:

  1. Absolute neutrophil count ≥1.5×109/L, platelet ≥100×109/L, hemoglobin ≥9g/dL;
  2. Bilirubin ≤ 1.5 times ULN (patients drained by retrograde technique may be included); ALT and AST ≤ 5 times ULN;
  3. Creatinine <120 μmol/L, or MDRD creatinine clearance rate> 60 mL/min;
* Women of childbearing age must undergo a negative pregnancy test (βHCG) before starting treatment. Women and men of childbearing age (sexual relationships with women of childbearing age) must agree to use them effectively during treatment and 6 months after the last dose of treatment Contraceptive measures;
* Signature of patient information and informed consent.

Exclusion Criteria:

* Women who are pregnant or nursing, or have fertility but refuse to take contraceptive measures;
* During the enrollment period, a serious active infection requiring antibiotic intravenous treatment occurred;
* Those who are allergic to test drugs;
* Presence of ≥2 grade neuropathy (CTCAE 5.0);
* Uncontrolled, symptomatic brain metastases or those with a history of difficult-to-control mental illness or severe intellectual or cognitive dysfunction;
* Suffering from active, known or suspected autoimmune diseases (including but not limited to: uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, vasculitis, hyperthyroidism, hypothyroidism and the need for bronchodilators Treatment of asthma, etc.). Subjects with hypothyroidism who only need hormone replacement therapy and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss) can be selected;
* Have been vaccinated or will be vaccinated with live vaccine within 30 days before the administration of Camrelizumab;
* Congestive heart failure, uncontrolled arrhythmia, myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months; or other patients who cannot tolerate surgery;
* Suffering from other malignant tumors within 5 years, except for fully treated cervical carcinoma in situ or squamous cell carcinoma of the skin, or basal cell carcinoma of the skin that has been basically controlled;
* Patients who cannot comply with the trial protocol or cannot cooperate with follow-up;
* The patient has already participated in another clinical trial;
* People deprived of their liberty or guardianship;
* Unable to receive medical supervision during the trial due to geographical, social or psychological reasons;
* Patients who cannot follow the trial protocol or cannot cooperate with follow-up;
* The researchers believe that it is not appropriate to participate in this experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | From date of starting treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  6-month progression-free survival rate

SECONDARY OUTCOMES:
ORR | From the first drug administration up to two years
  Overall Response Rate
DCR | From the first drug administration up to two years
  Disease Control Rate
PFS | From the first drug administration up to two years
  Progression Free Survival
Incidence of Treatment-Emergent Adverse Events | from the first drug administration to within 90 days for the last Camrelizumab combined with ablation and chemotherapy
  adverse events/serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, PhD, Principal Investigator — Harbin Medical University Cancer Hosptital